CLINICAL TRIAL: NCT03291327
Title: Evaluation of Two Active Lactobacilli for the Maintenance of Gingival Health: Double-Blind, Randomised Placebo-controlled Trial in Young Healthy Adults - a Proof of Principle Study
Brief Title: Evaluation of Two Active Lactobacilli for the Maintenance of Gingival Health
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to recruitment issues
Sponsor: Queen Mary University of London (Other)
Collaborators: Symrise AG (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QMERC2017/36
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2017-08

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Single Centre parallel arm (3) double blind placebo controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study randomisation schedule will be provided by an independent statistician in a sealed envelope and will be kept in a Study Master File (Test Products). The study blind will only be broken in an emergency where it was essential to know which formulation a participant had received in order to give the appropriate medical care. In the event of the requirement to break the code, the investigator (or designee) will, where possible, contact the Sponsor prior to breaking the blind. The investigator will then sign and date the broken code envelope and document the reason for breaking the code.
  All study products will be provided by the Sponsor, in blister packs pre-labelled with randomisation numbers according the Sponsor's randomisation schedule. Toothpaste with Fluoride (Colgate/Crest) together will also be provided.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Investigational product (Lactobacillus A) (Active Comparator): All volunteers considered to be suitable for the study will receive a pre-baseline dental prophylaxis. At baseline (BL) they will be instructed to abstain from all methods of tooth cleaning in mandible for 2 weeks (2W) apart from the fluoride toothpaste provided. A soft gum shield provided will cover the mandibular teeth whilst brushing and will be removed 10 minutes after brushing. Gingival health assessments and gingival crevicular fluid (GCF) and bacterial plaque samples be undertaken at BL and 2W. At 2W, all participants will receive a dental prophylaxis following the collection of samples and will be asked to resume their normal oral hygiene regime.
  Lactobacillus (A) in the form of a lozenge to be taken twice daily (in the morning and in the evening). The lactobacilli will be in the form of a lozenge, which should be placed on the tongue and allowed to dissolve. Any undissolved particles may be swallowed by the participant.
  Interventions: Dietary Supplement: Probiotics
- Investigational product (Lactobacillus B) (Active Comparator): All volunteers considered to be suitable for the study will receive a pre-baseline dental prophylaxis. At baseline (BL) they will be instructed to abstain from all methods of tooth cleaning in mandible for 2 weeks (2W) apart from the fluoride toothpaste provided. A soft gum shield provided will cover the mandibular teeth whilst brushing and will be removed 10 minutes after brushing. Gingival health assessments and gingival crevicular fluid (GCF) and bacterial plaque samples be undertaken at BL and 2W. At 2W, all participants will receive a dental prophylaxis following the collection of samples and will be asked to resume their normal oral hygiene regime.
  Lactobacillus (B) in the form of a lozenge to be taken twice daily (in the morning and in the evening). The lactobacilli will be in the form of a lozenge, which should be placed on the tongue and allowed to dissolve. Any undissolved particles may be swallowed by the participant.
  Interventions: Dietary Supplement: Probiotics
- Placebo Product (P) (Placebo Comparator): All volunteers considered to be suitable for the study will receive a pre-baseline dental prophylaxis. At baseline (BL) they will be instructed to abstain from all methods of tooth cleaning in mandible for 2 weeks (2W) apart from the fluoride toothpaste provided. A soft gum shield provided will cover the mandibular teeth whilst brushing and will be removed 10 minutes after brushing. Gingival health assessments and gingival crevicular fluid (GCF) and bacterial plaque samples be undertaken at BL and 2W. At 2W, all participants will receive a dental prophylaxis following the collection of samples and will be asked to resume their normal oral hygiene regime.
  Placebo (P) in the form of a lozenge to be taken twice daily (in the morning and in the evening). The placebo will be in the form of a lozenge, which should be placed on the tongue and allowed to dissolve. Any undissolved particles may be swallowed by the participant.
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — Lozenges for Home use

SUMMARY:
The objective of the study will be to demonstrate the effects of two active lactobacilli (A/B) and determine whether there are any changes in plaque accumulation, gingival health, immunological and microbial markers compared to a placebo (P) over a 2-week period of refraining from normal oral hygiene practice. This is a single centre, randomised, double-blind, parallel group study (3-Arm) of healthy subjects aged 18-30 years designed to demonstrate the effectiveness of two active lactobacilli using the experimental gingivitis Model: A proof of principle study on plaque, gingival status, immunological and microbial markers compared to placebo.

DETAILED DESCRIPTION:
This is a single centre, randomised, double-blind, parallel group study (3-Arm) of healthy subjects aged 18-30 years designed to demonstrate whether two active lactobacilli in the Experimental Gingivitis Model modify plaque accumulation, gingival status, immunological and microbial markers compared to placebo. Participants will be screened at a pre-baseline visit by a Study Dentist to determine their suitability for the study which will include healthy volunteers and exclude subjects with initial signs of gingival inflammation. Those volunteers considered to be suitable for the study will receive a pre-baseline dental prophylaxis. Participants will be required to return to the Study Centre 14 days following the screening visit and volunteers who comply with all the inclusion and exclusion criteria will be randomly allocated to one of three treatment groups at the baseline visit. Two of the groups will receive one of two probiotics containing either Lactobacillus (A) or Lactobacillus (B). The third group will receive placebo (P) which does not contain any active ingredient. Each subject will receive a fluoride toothpaste (Colgate Regular) and toothbrush (Oral-B) at the pre-baseline visit to reduce any carry-over (anti-microbial) effects from their normal toothpaste usage.

The initial brushing with the gum shield in place will be conducted under supervision by the study staff at the study centre to enable participants to be familiar with using the gum shield during their unsupervised brushing at home. Each participant will be given both verbal and written instructions, to enable them to correctly insert the gum shield under supervision; the placement of the gum shield will be checked by a study staff member, followed by supervised brushing of the upper teeth.

At the baseline visit those participants who fulfil the inclusion/exclusion criteria will receive a fluoride toothpaste (Colgate Regular) and toothbrush (Oral-B) for use throughout the duration of the study. All treatments will be unsupervised at the subject's home. Participants will be provided with a participant diary at the screening visit to check for compliance with tooth brushing throughout the study period. At the baseline visit those volunteers who successfully completed the inclusion/exclusion criteria will continue to complete the participant diary for compliance with twice daily tooth brushing, the test and control products and the placement of the gum shield over the lower teeth when brushing the upper teeth during the study. Those participants who fail to satisfy the inclusion/exclusion criteria will return the diary together with the fluoride toothpaste and toothbrush at the baseline visit.

Participants will be instructed to abstain from all methods of tooth cleaning in the lower (mandible) jaw for two weeks apart from the fluoride toothpaste provided by the study centre. A soft acrylic stent (gum shield) will be fabricated to cover the teeth in the lower jaw (mandible) whilst brushing the teeth in the upper (maxilla) jaw and will be removed 10 minutes after brushing. The soft stent can be easily inserted and removed without disturbance of the developing plaque whilst ensuring participants do not brush their lower teeth and thus disrupt plaque formation. Modified Gingival Index (MGI) (Lobene et al. 1986) assessments will be undertaken prior to the other assessments as this is non-invasive assessment. At baseline and after two weeks (+ 14 days) four sites/tooth (mesial, mid-buccal, distal and lingual) will be probed using the Gingival Bleeding Index [GBI]) as defined by Saxton & van der Ouderaa (1989) to assess the health status of the gingiva. Probing following one week of plaque accumulation will be avoided as bleeding in the gingival crevice may influence the developing biofilm. Non-invasive samples of gingival crevicular fluid (GCF) will however, be collected at all-time intervals before the BOP measurements or plaque sampling as the volume of GCF (Kistler et al. 2013) has been shown to increase before the development of clinically evident inflammation e.g. GBI. The GCF samples will be collected from the mesio-buccal sites of 4 selected sites (two teeth in each quadrant of the lower [mandible] jaw) on perio strips (ProFlow Inc. Amityville, NY) (Thunell et al. 2010). The strip will be applied in the gingival sulcus for 30 seconds to collect a standardised GCF fluid sample. The GCF samples will be pooled from 4 sites of each participant as indicated above at each time point and analysed on an individual basis. The number of sites with clearly visible plaque following the disclosing of the teeth in the lower (mandible) jaw (modified Quigley-Hein) (Turesky et al. 1970) will be recorded. Plaque will be collected from the buccal and lingual surfaces of teeth in the lower (mandible) jaw excluding 3rd molars from each participant using a sterile curette and placed in tubes with saturated saline-DMSO buffer. The plaque samples, and GCF samples in tubes with Phosphate Buffered Saline (PBS), will be transported on dry ice and stored at -80°C. All assessments and sample collection will be undertaken by trained and calibrated personnel. After two weeks, all participants who complete the study will receive a dental prophylaxis following the collection of samples and will be asked to resume their normal oral hygiene regime.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
2. Age Aged 18-30 years.
3. Compliance Understands and is willing, able and likely to comply with all study procedures and restrictions.
4. General Health Healthy volunteer

   Good general and mental health, in the opinion of the investigator or medically qualified designee:

   No clinically significant and relevant abnormalities of medical history or physical and oral examination.

   Absence of any condition that would impact on the subject's safety, or wellbeing, or affect the individual's ability to understand the study procedures and requirements.
5. Contraception Females of childbearing potential who are, in the opinion of the investigator, practising a reliable method of contraception. To exclude any confounding effects of pregnancy related changes in dental health. Adequate contraception is defined as abstinence, oral contraceptive, either combined or progestogen alone OR injectable progestogen OR implants of levonorgestrel OR estrogenic vaginal ring OR percutaneous contraceptive patches OR intrauterine device or intrauterine system OR double barrier method (condom or occlusive cap [diaphragm or cervical vault caps] plus spermicidal agent [foam, gel, film, cream, suppository]) OR male partner sterilization prior to the female subject's entry into the study, and this male is the sole partner for that subject. Following consent, Females will be required to use a pregnancy test kit administered at the study centre at Visit 1, results will be recorded on the relevant Case Report Form (CRF) and treated in confidence.
6. Dental Requirements At least eight teeth in the lower jaw with a minimum of 4 teeth in each quadrant BPE scores 0-2 in the lower (mandible) jaw Bleeding Score of <15% of sites in the lower (mandible) jaw (BOP) Following the dental prophylaxis, participants should have little or no gingival inflammation (<1) in the lower (mandible) jaw as assessed by MGI.
7. General Requirement Agree not to consume any other probiotic or yoghurt products during the study. Agree not to chew chewing gum during the study.

Exclusion Criteria:

1. Any inclusion criteria not met
2. Any disease which in the investigator's opinion could affect the participant's response to treatment, including in particular:

   * Diabetes mellitus Type I and II
   * Presence or recent history of infectious diseases such as AIDS, Hepatitis and tuberculosis or other respiratory infections including those that can be transmitted in saliva.
   * Bronchitis, tonsillitis or sinusitis.
3. Substance abuse e.g. smoking or chewing of tobacco or paan, drugs and alcoholism. E-cigarettes will also be excluded
4. Recent use of antibiotics and/or anti-inflammatory medication (within 4 weeks of visit).
5. Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.
6. Allergy/Intolerance to the test and placebo products (ingredients) in particular lactose and milk protein content (allergens) in the test products.
7. Evidence of chronic periodontitis (BPE score >3 in any sextant of the lower jaw)
8. Bleeding Score of >15% of sites in the lower (mandible) jaw
9. MGI Score of >1 (mean) in the lower (mandible) jaw
10. Currently ongoing treatment for chronic periodontitis
11. Currently using an anti-microbial mouth rinse
12. Participation in another clinical study or receipt of an investigational drug within 60 days of the screening visit.
13. Previous participation in this study.
14. Clinical dental students (2-5 years) will be excluded.
15. Ongoing or planned elective dental treatment involving endodontic treatment and crown and bridge preparation.

Furthermore, any participant requiring to undergo any emergency dental treatment during the study period will be assessed to determine whether they should continue to participate or be excluded.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Changes in gingival health status as indicated by changes in Gingival Bleeding Index (GBI) | Baseline to +14 days
  Changes in the gingival health status following the application of each test product will be performed using validated tools namely bleeding on probing (GBI) on test group subjects compared to placebo subjects.
  The presence or absence of bleeding will be scored within 30 seconds after probing with a Williams periodontal probe.
  Score Description 0 Absence of bleeding after 30 seconds.
  1. Bleeding observed after 30 seconds.
  2. Immediate bleeding observed.
Changes in gingival health status as indicated by changes in Quigley-Hein Plaque Index (Q-H) | Baseline to +14 days
  Changes in the gingival health status following the application of each test product will be performed using assessment of plaque accumulation (Q-H) on test group subjects compared to placebo subjects.
  All teeth in mandible excluding third molars will be scored with Quigley-Hein Plaque Index (Q-H).
  The teeth will be lightly dried a disclosing solution (PlaqueSearch TePe® TePe Munhygienprodukter, Malmo, Sweden) will be applied to all teeth in the mandible jaw. All teeth in the lower (mandible) jaw excluding 3rd molars will be visually scored using the Index, both buccal and lingual aspects of each tooth will be assessed.
  Score Description 0 No plaque.
  1. Isolated areas of plaque at gingival margin.
  2. Thin band of plaque at gingival margin (< 1mm).
  3. Plaque covering up to 1/3 of tooth surface.
  4. Plaque covering 1/3 to 2/3 of tooth surface.
  5. Plaque covering > 2/3 of tooth surface.
Changes in gingival health status as indicated by changes in Modified Gingival Index (MGI) | Baseline to +14 days
  Changes in the gingival health status following the application of each test product will be performed using colour changes in the gingiva (MGI) of test group subjects compared to placebo subjects.
  All teeth in mandible excluding third molars will be scored with MGI Score Description 0 Absence of inflammation.
  1. Mild inflammation; slight change in colour, little change in texture of any portion of but not the entire marginal or papillary gingival unit.
  2. Mild inflammation; criteria as above but involving the entire marginal or papillary gingival unit.
  3. Moderate inflammation; glazing, redness, oedema, and/or hypertrophy of the marginal or papillary gingival unit.
  4. Severe inflammation; marked redness, oedema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion or ulceration.

SECONDARY OUTCOMES:
Changes in Inflammatory Markers | Baseline to + 14 days
  To assess changes in inflammatory markers in Gingival Crevicular Fluid following use of each test product
Changes in Bacterial Composition | Baseline to + 14 days
  To assess changes in bacterial composition in collected plaque samples following use of each test product

IPD SHARING:
Plan to Share IPD: No